CLINICAL TRIAL: NCT06788847
Title: Advancing Dupuytren's Contracture Treatment: a Clinical Prospective Study on Ultrasound-Guided Needle Knife Dissection
Brief Title: Evaluating Ultrasound-Guided Needle Knife for Dupuytren's Contracture
Acronym: DC-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Maher Ismail Ahmed Elashmawy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Maher Ismail Ahmed Elashmawy, Lecturer of Rheumatology, Physical Medicine and Rehabilitation, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MansouraUH_DC-US_2025; R.24.12.2966 (Registry Identifier: Mansoura University Faculty of Medicine IRB)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Dupuytren Contracture
Keywords: Ultrasound-Guided Procedure; Dupuytrene's Contracture; Tubiana Grade; Fibrotic Cords Acupotomy; Functional Hand Recovery; Palmar Fascia Fibrosis
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Intervention Model Description: All participants will undergo ultrasound-guided needle knife dissection for Dupuytren's Contracture treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group: Ultrasound-Guided Needle Knife Dissection (Experimental): Participants in this group will undergo ultrasound-guided needle knife dissection for the treatment of Dupuytren's Contracture. Local anesthesia using 3-5ml of 1% lidocaine 0.25% bupivacaine is administered for patient comfort. This procedure is designed to improve hand function with minimal complications.
  Interventions: Procedure: Ultrasound guided needle knife dissection

INTERVENTIONS:
Procedure: Ultrasound guided needle knife dissection — This procedure involves a minimally invasive dissection of the fibrous cords in Dupuytren's Contracture using a needle knife guided by ultrasound imaging. Local anesthesia using 3-5 ml of 1% Lidocaine and 0.25% bupivacaine is administered for patient comfort. The technique aims to improve precision, minimize complications and reduce recurrence.
  Device: Sonosite M-Turbo Ultrasound Machine with Linear Probe HFL38x (6-13 MHz) is used for real-time imaging during the procedure.
  Other Names: UGNK procedure

SUMMARY:
This study aims to evaluate the efficacy and safety of ultrasound-guided needle knife dissection in treating Dupuytren's contracture. The procedure is designed to improve hund function and minimize complications associated with the conventional surgical methods.

DETAILED DESCRIPTION:
Dupuytren's contracture is a disease mainly characterized by the progressive fibrosis of the palmar fascia with subsequent hand deformity and dysfunction. The current study seeks to explore, through this minimally invasive technique, ultrasound-guided needle knife dissection regarding ROM and patient satisfaction. The procedure will be carried out under ultrasound guidance to ensure safety and completeness with the accuracy of precise dissection. Primary outcome measures will concern hand mobility, and secondary measures will evaluate patient self-reported satisfaction and any complications for the 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Dupuytren's Contracture.
* Willing to undergo ultrasound-guided needle knife dissection

Exclusion Criteria:

* Patients who have undergone previous surgery or needle apponeurotomy for Dupuytren's Contracture on the same hand.
* Active hand infections, open wounds, or dermatological conditions in the treatment area.
* Coagulopathy or use of anticoagulant that cannot be safely paused
* Neuromuscular disorders affecting hand function
* Pregnancy or breastfeeding
* Uncontrolled systemic illnesses, such as poorly managed diabetes or cardiovascular disease.
* Known hypersensitivity to local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Improvement in hand Function | 6 months
  Functional Improvement:
  - Evaluated using the QuickDASH score (0-100 scale).
Improvement in hand mobility | 6 months
  Range of Motion (ROM):
  - Measurment of joint mobility in degrees at MCP and PIP joints by goniometer.

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  Evaluation of patient-reported satisfaction using a standardized questionnaire.
Rate of procedure-related complications | 6 months
  Monitoring and documentation of procedure-related complications, including infection, nerve injury, and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared to ensure participant confidentiality and comply with ethical and institutional regulations. The collected data will only be used for the purposes of this study and will not be disclosed to external parties